CLINICAL TRIAL: NCT02779621
Title: A Pragmatic Randomized Control Trial Which Evaluates the Potential for HPV Self-testing to Promote Participation in Cervical Screening (PROMOTER) Trial
Brief Title: The Potential for HPV Self-testing to Promote Participation in Cervical Screening
Acronym: PROMOTER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Chief Investigator relocating out of the United Kingdom.
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Abbott (Industry); Copan Italia SPA , Via F. Perotti, 10, 25125 Brescia, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 203560
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Cervix Diseases
MeSH Terms: conditions — Uterine Cervical Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-sampling (Experimental): (Self-collecting a vaginal sample with a swab for HPV testing) Women in the experimental arm will have the option of vaginal self-sampling for HPV testing, in addition to the routine screening test. They can choose one of them.
  Interventions: Procedure: Self-collecting a vaginal sample with a swab for HPV testing; Procedure: Collection of cervical sample for routine cervical screening
- Routine smear (Active Comparator): (Collection of cervical sample for routine cervical screening) Women in the control arm will only receive the routine cervical screening invitation letter.
  Interventions: Procedure: Collection of cervical sample for routine cervical screening

INTERVENTIONS:
Procedure: Self-collecting a vaginal sample with a swab for HPV testing — The vaginal sample self-collected with the Floq swab will be tested for Human Papillomavirus (HPV) using Abbott RealTime PCR assay.
  Other Names: Copan Floq is used for self-sampling
  Arms: Self-sampling
Procedure: Collection of cervical sample for routine cervical screening — This is the routine cervical screening test available to the public through the NHS. This sample is collected by a clinician (usually a Practice Nurse)
  Other Names: Routine cervical smear test

SUMMARY:
To explore the potential for vaginal self-sampling to increase participation in cervical screening, we offer the option of self-sampling to a group of non-participants in cervical screening (intervention), in addition to the routine screening (smear) test. Women in the control group will only receive the routine screening invitation letter. The total screening uptake rate, 2 months since the recruitment in each group will be compared.

DETAILED DESCRIPTION:
The aim of this research is to assess the feasibility of making vaginal self sampling available to women who have declined smear testing (defaulters), through the NHS to prevent cervical cancer. We plan to identify all defaulters living in Coventry between 30 and 40 years (n≈6000) from the cervical screening call-recall system. They will be randomized 1:1 to intervention and control arms. Women in the control arm will be sent a routine screening letter reminding them to have a smear test. Women in the intervention arm will be given the option of self-sampling for HPV testing, if they do not wish to have a smear test. They could order a self-HPV test by returning a slip in the pre-paid envelope. We then send the woman a vaginal self-collection kit. Self-collected sample will be returned to the laboratory for HPV testing. Whilst HPV positives (10-15%) will be advised to have a smear test, HPV negatives will be advised to accept their next smear test invitation.

ELIGIBILITY:
Inclusion Criteria:

* All cervical screening programme defaulters living in Coventry

Exclusion Criteria:

1. Pregnancy
2. Total hysterectomy (abdominal/laparoscopic/vaginal)
3. Never been sexually active/ intimate
4. Women who cannot give valid, informed, written consent
5. HPV self-sample returned without a signed consent form
6. Women who request the research team to be excluded from the trial
7. Women who have written to the Screening Services to record their refusal to take part in the NHSCSP
8. Women who are identified as becoming pregnant or undergoing hysterectomy following the initial test will be excluded from the analysis of data for secondary outcomes

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Estimated); Primary Completion 2017-01 (Estimated); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
The total screening uptake rate in each arm | 2 months since the recruitment
  In the experimental arm, the numerator will be the total number of smear tests + HPV self-tests. In the active control arm, it will be total number of smear tests.

SECONDARY OUTCOMES:
Proportion of HPV positive women who have subsequently had a smear test | 2 months since the HPV test result
Proportion of smear positive women referred to colposcopy | 1 month since the smear result
Proportion of women referred to colposcopy had attended colposcopy | 3 months since the smear result
Proportion of women attended colposcopy had a CIN2+ | 4 months since the smear result
Assess the women's attitude towards self-sampling and its feasibility | 2 months since the recruitment
  Analysing data of user questionnaires
Assess the women's attitude towards the feasibility of self-sampling | 2 months since the recruitment
  Analysing data of user questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ceri Jones, Study Director — Head of Research, Development & Innovation, UHCW, Coventry
Locations (1):
- University Hospital of Coventry & Warwickshire, Coventry, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No